CLINICAL TRIAL: NCT01485354
Title: The Effect of Repetitive Upper Arm Training in a Virtual Environment on Upper Extremity Motor Recovery in Chronic-stroke Survivors
Brief Title: Upper Arm Training With Armeo Spring for Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001255
Record Dates: First submitted 2011-06-28; First posted 2011-12-05 (Estimated); Results first posted 2017-07-12 (Actual); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Armeo Spring training (Experimental): Subjects will participate in upper extremity rehabilitation using the Armeo Spring system for a period of 6 weeks. The intervention will consist of 18 training sessions (60 minute sessions, 3 times a week).
  Interventions: Device: Armeo Spring training

INTERVENTIONS:
Device: Armeo Spring training — Upper-limb training using the Armeo system for a period of 6 weeks
  Other Names: Armeo Spring (Hocoma AG, Switzerland)

SUMMARY:
The purpose of this study is to assess the clinical outcomes of upper extremity training using the Armeo Spring system in a chronic post-stroke population with impaired upper extremity function.

DETAILED DESCRIPTION:
The Armeo Spring system is an adjustable arm orthosis that has received FDA 510K clearance. It passively counterbalances the weight of the arm, thereby reducing the effort required to overcome gravity during the performance of upper-limb movements. The device provides subjects with augmented feedback via a virtual environment (i.e. computer games). The tasks to be performed in the virtual environment are designed to achieve functional movements, such as arm reaching movements.

The goal of the study is to assess the clinical outcomes of upper extremity training using the Armeo Spring system in a chronic post-stroke population with impaired upper extremity function. The Armeo Spring system is equipped with a grip sensor that subjects squeeze with their hand to interact with virtual objects during the games. In a first phase of the study, we attempted to replace the grip sensor that is part of the system with a sensorized glove, to facilitate a more natural movement of hand opening/closing. However, we experienced technical difficulties with the sensorized glove and decided to abandon this aim for the purpose of gathering data about the clinical outcomes of upper extremity training using the Armeo Spring system.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, community dwelling, age 18-70
* First-time non-traumatic ischemic or hemorrhagic stroke at least 3 months prior to study enrollment
* Score of 15-55 out of 66 on arm motor Fugl-Meyer scale
* The ability to extend >=10 degrees at metacarpophalangeal and interphalangeal joint of all digits

Exclusion Criteria:

* Cognitive impairment that may interfere with understanding instructions for motor tasks and assessment tools
* Inability to operate the Armeo system (subjects must have sufficient range of movement to enable calibration of the virtual workspace)
* Participation in other forms of therapy/intervention for upper extremity motor recovery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited primarily among the outpatient population of stroke survivors at Spaulding Rehabilitation Hospital. We primarily relied upon a registry of stroke survivors who had agreed to be contacted for research studies with focus on stroke rehabilitation.
Groups:
- Armeo Spring Training: Subjects participated in upper extremity rehabilitation using the Armeo Spring system for a period of 6 weeks. The intervention consisted of 18 training sessions (60 minute sessions, 3 times a week).
  Armeo Spring training: Upper-limb training using the Armeo system for a period of 6 weeks
Period: Overall Study
Arm/Group | Armeo Spring Training
Started | 17
Completed | 12
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Upper-extremity Fugl-Meyer Score (Measure of Motor Impairment) (i.e. Difference Between Fugl-Meyer Score at Baseline and at Completion of the 3-week Intervention)
Description: The upper-extremity Fugl-Meyer scale allow one to assess the severity of motor impairments in stroke survivors using a scale from 0 (severe impairment) to 66 (no impairment). It is based on visual observations gathered by asking subjects to perform upper-limb movements using the stroke-affected limb. Therapists rate the performance of the motor tasks using an ordinal scale ranging from 0 (cannot perform) to 2 (can perform fully) that captures the motor ability of the individual. The investigators computed the difference between the Fugl-Meyer score at completion of the 3-week intervention and the Fugl-Meyer score at baseline.
Time Frame: Data collected at baseline and at completion of the 3-week intervention
Population: Please notice that we recruited 17 subjects, but 5 subjects withdrew from the study. Herein, we report the results for those subjects who completed the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 12
units on a scale | 6.4 (6.0)

2. Secondary Outcome: Change in Wolf Motor Function Test Score (a Functional Test) (i.e. Difference Between Wolf Motor Function Test Score at Baseline and at Completion of the 3-week Intervention)
Description: The Wolf Motor Function test is designed to assess the severity of functional limitations in stroke survivors. The scale is administered by asking subjects to perform a series of functional movements (e.g. reach for and pick up a paperclip). The outcome of the assessment is the average time needed to perform the motor tasks that are part of the assessment. The score ranges from 0 to 120 s (i.e. if the subject is unable to perform the task, the score for that task is set to 120 s). The investigators computed the difference between the Wolf Motor Function Test score at completion of the 3-week intervention and the Wolf Motor Function Test score at baseline.
Time Frame: Data collected at baseline and at completion of the 3-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 12
sec | 6.6 (12.6)

3. Secondary Outcome: Change in Functional Ability Scale Score (Scale to Rate Quality of Movement) (i.e. Difference Between Functional Ability Scale Score at Baseline and at Completion of the 3-week Intervention)
Description: The Functional Ability Scale is designed to assess the quality of movement during the performance of a battery of functional tasks. Therapists observe the subject while performing the motor tasks and use an ordinal scale to rate the quality of movement. The scale used to rate each motor task ranges from 0 to 5. The Functional Ability Scale is derived by adding up the scores for each motor task performed by the subject. Subjects perform 15 motor tasks. Hence the Functional Ability Scale score varies from 0 (very poor quality of movement) to 75 (physiological movement). The investigators computed the difference between the Functional Ability Scale score at completion of the 3-week intervention and the Functional Ability Scale score at baseline.
Time Frame: Data collected at baseline and at completion of the 3-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 12
units on a scale | 0.3 (0.6)

4. Secondary Outcome: Change in Box and Block Test Score (Manual Dexterity Test) (i.e. Difference Between Box and Block Test Score at Baseline and at Completion of the 3-week Intervention)
Description: The Box and Block test is designed to assess manual dexterity in subjects with motor impairments. Subjects are asked to move small wooden blocks from one box to another, moving their stroke-affected arm over a divider between the two boxes. The output of the test is the number of blocks that the subject moves from one box to the other within a set amount of time (i.e. 1 min). Older adults who are otherwise healthy would typically move 60 to 70 blocks in 1 min. Hence, the range of the scale for older adults is 0 to 70. The investigators computed the difference between the Box and Block Test score at completion of the 3-week intervention and the Box and Block Test score at baseline.
Time Frame: Data collected at baseline and at completion of the 3-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of blocks
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 12
number of blocks | 1.1 (3.2)

5. Secondary Outcome: Change in Grip Strength (Strength Test) (i.e. Difference Between Grip Strength at Baseline and at Completion of the 3-week Intervention)
Description: This test is carried out by using a hand dynamometer that measures the grip strength of the individual in kilograms (used as a measure of force). Subjects are instructed to position the thumb on one handle of the dynamometer and the other fingers on the other handle of the dynamometer. The device measures the force generated by the subject using a power grip. The investigators computed the difference between the Grip Strength value at completion of the 3-week intervention and the Grip Strength value at baseline.
Time Frame: Data collected at baseline and at completion of the 3-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Armeo Spring Training
Number analyzed (Participants) | 12
kg | 3.0 (5.2)

ADVERSE EVENTS:
Time Frame: We collected information in regard to potential adverse events during the 3 weeks of the study intervention.
Arm/Group | Armeo Spring Training
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No